CLINICAL TRIAL: NCT05387460
Title: Radiomics Based on Multimodal Transvaginal Ultrasound Imaging in Predicting Endometrial Cancer and Cervical Stromal Invasion
Brief Title: Radiomics Based Multimodal Transvaginal Ultrasound Imaging in Endometrial Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Tongji Hospital (Other)
Collaborators: Women's Hospital School Of Medicine Zhejiang University (Other)
Responsible Party: Principal Investigator, Qinglei Gao, Professor, Tongji Hospital
Other Study IDs: 2022-TJ-R-RBM
Record Dates: First submitted 2022-05-18; First posted 2022-05-24 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Endometrial Cancer; Cervical Stromal Invasion; Transvaginal Ultrasound
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Radiomics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Training cohort: The cohort of Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology is a training cohort Intervention/treatment
  Interventions: Diagnostic Test: radiomics
- validation cohort: The cohort of Women's Hospital, School of Medicine, Zhejiang University is a validation cohort
  Interventions: Diagnostic Test: radiomics

INTERVENTIONS:
Diagnostic Test: radiomics — Radiomics refers to high-throughput mining of quantitative image features from medical imaging. Radiomics derived data, when combined with other pertinent clinicopathological features, can produce accurate and robust evidence-based decision-making systems. Multimodal radiomics can provide more imaging feature information than single modal radiomics, which showed better diagnostic performance in previous study of kinds of cancer diseases.

SUMMARY:
Retrospectively collect preoperative transvaginal B-mode ultrasound (BMUS), color Doppler flow imaging (CDFI) and three-dimensional ultrasound (3D-US) images and clinical data in patients with non-endometrial cancer diseases and endometrial cancer confirmed by pathology. They were grouped as training set(Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology) and external validation set(Women's Hospital, School of Medicine, Zhejiang University) . Radiomics features were extracted from corresponding transvaginal ultrasound images. Then, the minimum redundancy maximum relevance (mRMR) algorithm and the least absolute shrinkage and selection operator (LASSO) regression were used to select the non- malignant or malignant status-related features and cervical stromal invasion (CSI) status or non-CSI status features and construct the transvaginal ultrasound radiomics score (Rad-score). Multivariate logistic regression was performed using the three radiomics score together with clinical data, and subsequently develop a nomogram to diagnosis endometrial cancer and CSI respectively. The performance of the nomogram was assessed by discrimination, calibration, and clinical usefulness in the training and external validation set.

DETAILED DESCRIPTION:
Endometrial Cancer is the second most common gynecological cancer in China and the first in Western countries. The common clinical symptom of endometrial cancer is vaginal bleeding, which occurs in about 10% of postmenopausal women. Most patients with postmenopausal vaginal bleeding are diagnosed with benign diseases, and less than 10% of patients are diagnosed with endometrial cancer. Early diagnosis is crucial for the prognosis of patients with endometrial cancer. The 5-year survival rate of patients with endometrial cancer which lesions localized to the uterus is about 95%, while the survival rate of patients with regional and distant metastasis is reduced to less than 70% and 20%.

Surgery is the main treatment of endometrial cancer. CSI is one of the main criteria for determining the follow-up treatment. According to NCCN guidelines, Total Hysterectomy and Bilateral Salpingo-Oophorectomy (THBSO) are standard treatments for patients with endometrioid carcinoma without CSI. While extensive hysterectomy or surgery after radiotherapy is appropriate for patients with CSI. Therefore, accurate assessment of CSI status in patients with EC before operation is important for the formulation of accurate surgical strategies.

Endometrial biopsy has been considered the gold standard for assessing endometrial cancer. However, it is limited because of increased cost, sample errors, related complications such as pain, bleeding, inability to evaluate the extent of tumor invasion and easy to cause tumor spread. CT/MR are alternative ways with high cost and complications. Transvaginal ultrasound examination is considered as the first imaging investigation for endometrial cancer. ESGO/ESTRO/ESP guidelines for the management of patients with endometrial carcinoma indicate that transvaginal ultrasound can be used instead of magnetic resonance imaging to detect cervical stromal infiltration under the operation of experienced doctors. Improving the performance of ultrasonic diagnosis is significant for how to choose the follow-up treatment and reduce the cost and risk of overtreatment.

Radiomics refers to high-throughput mining of quantitative image features from medical imaging. Radiomics derived data, when combined with other pertinent clinicopathological features, can produce accurate and robust evidence-based decision-making systems. Multimodal radiomics can provide more imaging feature information than single modal radiomics, which showed better diagnostic performance in previous study of kinds of cancer diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed by operation and pathology
2. Patients with preoperative transvaginal ultrasound images

Exclusion Criteria:

1. Past history of gynecological malignant tumors
2. Previous pelvic surgery or radiotherapy or chemotherapy
3. Poor image quality
4. Incomplete pathological or diagnosis report

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Endometrial cancer can only happen in females.
Study Population: Patients who had Endometrial cancer or benign endometrial diseases and completed the transvaginal ultrasound examination before operation
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
AUC value | through study completion, an average of 1 year
  Area under the receiver operating characteristic (ROC) curve (AUC）

SECONDARY OUTCOMES:
Diagnostic specificity | through study completion, an average of 1 year
  diagnosis specificity of intelligent ultrasound analysis
Diagnostic sensitivity | through study completion, an average of 1 year
  diagnosis sensitivity of intelligent ultrasound analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No